CLINICAL TRIAL: NCT00163098
Title: A Multi-Centre, Multinational, Randomized, Double-Blind, Placebo Controlled, Proof Of Concept Trial To Assess The Effects Of A Subject-Optimized Dose Of UK-369,003 On Exercise Capacity In Subjects With Chronic Obstructive Pulmonary Disease
Brief Title: A Study of UK-369,003 on the Safety and Efficacy in Patients With COPD
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A3711028
Record Dates: First submitted 2005-09-08; First posted 2005-09-13 (Estimated); Last update posted 2006-10-13 (Estimated); Status verified 2006-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — 1-(6-ethoxy-5-(3-ethyl-6,7-dihydro-2-(2-methoxyethyl)-7-oxo-2H-pyrazolo(4,3-d)pyrimidin-5-yl)-3-pyridyl sulphonyl)-4-ethylpiperazine

INTERVENTIONS:
Drug: UK-369,003

SUMMARY:
A randomised, controlled study investigating the effect of UK-369,003 on exercise tolerance in patients with COPD

ELIGIBILITY:
Inclusion Criteria:

* GOLD criteria 2 to 4
* 10 pack year history of smoking

Exclusion Criteria:

* Women of child bearing potential

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136
Dates: Start 2004-12; Study Completion 2005-12

PRIMARY OUTCOMES:
Effect on exercise tolerance

SECONDARY OUTCOMES:
Effect on lung function and quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (25):
- Argentina (8):
  - Pfizer Investigational Site, Córdoba, Córdoba Province
  - Pfizer Investigational Site, San Miguel de Tucumán, Pcia de Tucuman
  - Pfizer Investigational Site, Rosario, Santa FÃ©
  - Pfizer Investigational Site, Buenos Aires
  - Pfizer Investigational Site, Ciudad de Beurnos Aires
  - Pfizer Investigational Site, Ciudad de Buenos Aires,
  - Pfizer Investigational Site, Ciudad de Buenos Aires
  - Pfizer Investigational Site, Provincia de Buenos Aires
- Australia (6):
  - Pfizer Investigational Site, Camperdown, New South Wales
  - Pfizer Investigational Site, Darlinghurst, New South Wales
  - Pfizer Investigational Site, Chermside, Queensland
  - Pfizer Investigational Site, Adelaide, South Australia
  - Pfizer Investigational Site, Melbourne, Victoria
  - Pfizer Investigational Site, Perth, Western Australia
- Germany (2):
  - Pfizer Investigational Site, Giessen
  - Pfizer Investigational Site, Greifestein
- India (5):
  - Pfizer Investigational Site, Kochi, Kerala
  - Pfizer Investigational Site, Mumbai, Maharashtra
  - Pfizer Investigational Site, Pune, Maharashtra
  - Pfizer Investigational Site, Chennai, Tamil Nadu
  - Pfizer Investigational Site, Vellore, Tamil Nadu
- United Kingdom (3):
  - Pfizer Investigational Site, Papworth Everard, Cambridgeshire
  - Pfizer Investigational Site, Glasgow
  - Pfizer Investigational Site, Newcastle upon Tyne
- Pfizer Investigational Site

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3711028&StudyName=A+Study+of+UK%2D369%2C003+on+the+Safety+and+Efficacy+in+Patients+with+COPD+